CLINICAL TRIAL: NCT06742554
Title: Comparative Efficacy of Buprenorphine Transdermal Patch Versus Tramadol in Postoperative Analgesia for Shoulder Arthroscopy: a Randomized Controlled Trial.
Brief Title: Comparative Efficacy of Buprenorphine Transdermal Patch Versus Tramadol in Postoperative Analgesia for Shoulder Arthroscopy
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: medina medical center (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Salah Elsawy, Anesthesia and Pain Management Consultant, Director of Day Case Surgeries, medina medical center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BUT002/2024
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Pain; Shoulder Pain; Opioid Analgesia; Tramadol; Buprenorphine; Arthroscopy; Interscalene Brachial Plexus Block; Analgesic
Keywords: buprinorphin; transdermal; tramadol
MeSH Terms: conditions — Pain, Postoperative; Shoulder Pain | interventions — Tramadol

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-assignment study where participants are allocated to one of two intervention groups. Group A will receive a Buprenorphine 10 mg transdermal patch applied 4 hours prior to surgery, providing sustained analgesia for up to 72 hours postoperatively. Group B will receive Tramadol at a standard dosage (100 mg every 8 hours as needed for pain) starting postoperatively. Both groups will receive interscalene brachial plexus block (ISBPB) as part of their intraoperative anesthesia.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Buprenorphine Transdermal Patch (Active Comparator): Participants in this arm will receive a 10 mg Buprenorphine transdermal patch, applied 4 hours before shoulder arthroscopic surgery. The patch delivers a steady dose of Buprenorphine for up to 7 days, providing sustained postoperative analgesia. All participants will also undergo an interscalene brachial plexus block (ISBPB) as part of their anesthesia protocol.
  Interscalene Brachial Plexus Block: Administered intraoperatively using 25 mL of 0.5% bupivacaine.
  Interventions: Drug: Buprenorphine transdermal patch
- Tramadol (Active Comparator): Participants in this arm will receive Tramadol for postoperative pain management. The medication will be administered at a dose of 100 mg every 8 hours as needed, beginning after the interscalene brachial plexus block (ISBPB) wears off.
  Interscalene Brachial Plexus Block: Administered intraoperatively using 25 mL of 0.5% bupivacaine.
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Buprenorphine transdermal patch — Buprenorphine Transdermal Patch (10 mg): Applied once before surgery for continuous pain control.
  Interscalene Brachial Plexus Block: Administered intraoperatively using 25 mL of 0.5% bupivacaine.
  Arms: Buprenorphine Transdermal Patch
Drug: Tramadol — Tramadol: Administered orally or intravenously at a standard dose of 100 mg every 8 hours, based on patient-reported pain levels.
  Interscalene Brachial Plexus Block: Administered intraoperatively using 25 mL of 0.5% bupivacaine.
  Arms: Tramadol

SUMMARY:
This study compares the efficacy, safety, and patient satisfaction of the Buprenorphine 10 mg transdermal patch versus Tramadol for postoperative analgesia in shoulder arthroscopic surgery. The study hypothesizes that Buprenorphine provides superior pain relief with fewer side effects compared to Tramadol.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years.
* Patients undergoing elective shoulder arthroscopy.
* Classified as ASA (American Society of Anesthesiologists) physical status I or II.
* Able to provide informed consent.
* Willing to comply with study protocols and follow-up assessments

Exclusion Criteria:

* Known allergy or hypersensitivity to Buprenorphine, Tramadol, or any related compounds.
* History of substance abuse, opioid dependency, or chronic pain requiring ongoing analgesic therapy.
* Pregnant or breastfeeding individuals.
* Presence of severe hepatic, renal, or respiratory disease.
* Any psychiatric or neurological condition that might interfere with pain perception or reporting (e.g., dementia, severe anxiety).
* Participation in another clinical trial within the last 30 days.
* Inability to apply or tolerate a transdermal patch (e.g., due to skin disorders or sensitivities).
* Contraindications to interscalene brachial plexus block, such as infection at the site, coagulopathy, or pre-existing neuropathy in the upper limb.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain score | Pain intensity will be measured using the The numeric rating scale , recorded at 6, 12, 24, 48, and 72 hours after surgery.
  Postoperative pain scores measured using the The Numeric Rating Scale over 72 hours. It involves asking participants to rate their pain on a scale of 0 to 10, where:
  * 0 represents "No Pain"
  * 10 represents "Worst Possible Pain" Lower scores indicate better outcomes.
Duration of Effective Analgesia | From the time of surgery (Day 0) to 72 hours postoperatively.
  The time from the full recovery from the interscalene brachial plexus block (ISBPB) until 72 hrs postoperatively.

SECONDARY OUTCOMES:
Incidence of Adverse Effects | From the time of surgery (Day 0) to 72 hours postoperatively
  he number of participants experiencing adverse effects (e.g., nausea, vomiting, dizziness, sedation, or skin irritation) will be recorded. Data will be collected through direct patient reports and clinical observations.
Patient Satisfaction (Likert Scale) | At 72 hours postoperatively
  Patient satisfaction with pain management will be assessed using a 5-point Likert scale, where 1 indicates "very dissatisfied" and 5 indicates "very satisfied." Higher scores reflect better patient satisfaction
Early Mobilization and Rehabilitation Adherence | From 24 to 72 hours postoperatively.
  The ability to perform early mobilization and adhere to physiotherapy protocols (e.g., range-of-motion exercises) will be assessed by physical therapists. This will be rated as "Full adherence," "Partial adherence," or "No adherence." Full adherence indicates a better outcome.
Total Rescue Analgesic Consumption | From the time of surgery (Day 0) to 72 hours postoperatively
  The total amount of rescue analgesics (e.g., acetaminophen or additional opioids) required by each participant will be recorded in milligrams. Lower consumption indicates better efficacy of the primary analgesic.

CONTACTS AND LOCATIONS:
Locations (1):
- Medina Medical Center, Madinah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, including primary and secondary outcome measures, will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be made available upon publication of the study results in a peer-reviewed journal
Access Criteria: Researchers and healthcare professionals conducting methodologically sound and ethically approved research.
  Individuals or institutions with research objectives aligned with the scope of the study, such as meta-analyses or systematic reviews

REFERENCES:
- [Background] Arshad Z, Prakash R, Gautam S, Kumar S. Comparison between Transdermal Buprenorphine and Transdermal Fentanyl for Postoperative Pain Relief after Major Abdominal Surgeries. J Clin Diagn Res. 2015 Dec;9(12):UC01-4. doi: 10.7860/JCDR/2015/16327.6917. Epub 2015 Dec 1. PMID 26816973